CLINICAL TRIAL: NCT02786927
Title: An Open-label Study to Evaluate the Preference Attributes of the ELLIPTA™ Dry Powder Inhaler (DPI) Compared to the HandiHaler™ DPI in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Preference Attributes of ELLIPTA Dry Powder Inhaler (DPI) and HANDIHALER DPI in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 204983
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Results first posted 2017-06-22 (Actual); Last update posted 2018-10-15 (Actual); Status verified 2018-09

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: HANDIHALER; Dry Powder Inhaler; COPD; ELLIPTA; Inhaler preference attributes
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- ELLIPTA - HANDIHALER; HANDIHALER Questionnaire Version 1 (Experimental): Subjects will be dispensed the ELLIPTA inhaler at Visit 1 to use during the first period (once daily for 5-9 days), and the HANDIHALER inhaler at Visit 2 to use during the second period (once daily for 5-9 days). At Visit 3, subjects will complete Version 1 of the inhaler preference questionnaire.
  Interventions: Drug: Placebo ELLIPTA device; Drug: Placebo capsules for use in HANDIHALER device; Other: Inhaler Preference Questionnaire Version 1
- ELLIPTA - HANDIHALER; Questionnaire Version 2 (Experimental): Subjects will be dispensed the ELLIPTA inhaler at Visit 1 to use during the first period (once daily for 5-9 days), and the HANDIHALER inhaler at Visit 2 to use during the second period (once daily for 5-9 days). At Visit 3, subjects will complete Version 2 of the inhaler preference questionnaire.
  Interventions: Drug: Placebo ELLIPTA device; Drug: Placebo capsules for use in HANDIHALER device; Other: Inhaler Preference Questionnaire Version 2
- HANDIHALER - ELLIPTA; Questionnaire Version 1 (Experimental): Subjects will be dispensed the HANDIHALER inhaler at Visit 1 to use during the first period (once daily for 5-9 days), and the ELLIPTA inhaler at Visit 2 to use during the second period (once daily for 5-9 days). At Visit 3, subjects will complete Version 1 of the inhaler preference questionnaire.
  Interventions: Drug: Placebo ELLIPTA device; Drug: Placebo capsules for use in HANDIHALER device; Other: Inhaler Preference Questionnaire Version 1
- HANDIHALER - ELLIPTA; Questionnaire Version 2 (Experimental): Subjects will be dispensed the HANDIHALER inhaler at Visit 1 to use during the first period (once daily for 5-9 days), and the ELLIPTA inhaler at Visit 2 to use during the second period (once daily for 5-9 days). At Visit 3, subjects will complete Version 2 of the inhaler preference questionnaire.
  Interventions: Drug: Placebo ELLIPTA device; Drug: Placebo capsules for use in HANDIHALER device; Other: Inhaler Preference Questionnaire Version 2

INTERVENTIONS:
Drug: Placebo ELLIPTA device — Placebo ELLIPTA is a DPI device containing powder for inhalation, to be inhaled orally once daily for 5-9 days. It contains two strips with 30 blisters per strip - one strip contains lactose monohydrate whereas the other strip contains lactose monohydrate blended with magnesium stearate.
Drug: Placebo capsules for use in HANDIHALER device — Placebo capsules contain lactose monohydrate in the form of powder for inhalation, to be used with the HANDIHALER inhaler as an oral inhalation once daily for 5-9 days.
Other: Inhaler Preference Questionnaire Version 1 — Consists of 5 questions to assess subjects' preference of device attributes and dosing regimens. The two versions of the questionnaire ask the same questions, but differ in the ordering of inhalers in their responses.
  Arms: ELLIPTA - HANDIHALER; HANDIHALER Questionnaire Version 1; HANDIHALER - ELLIPTA; Questionnaire Version 1
Other: Inhaler Preference Questionnaire Version 2 — Consists of 5 questions to assess subjects' preference of device attributes and dosing regimens. The two versions of the questionnaire ask the same questions, but differ in the ordering of inhalers in their responses.
  Arms: ELLIPTA - HANDIHALER; Questionnaire Version 2; HANDIHALER - ELLIPTA; Questionnaire Version 2

SUMMARY:
This is a Phase IV multi-center, randomized, open-label, cross-over, placebo study in subjects with Chronic Obstructive Pulmonary Disease (COPD) to compare inhaler-specific preference attributes of two inhalers - ELLIPTA dry powder inhaler (DPI) and the HANDIHALER DPI. The primary objective of this study is to evaluate whether more subjects with COPD prefer the ELLIPTA inhaler to the HANDIHALER DPI based on the number of steps needed to take medication.

All subjects will use the ELLIPTA inhaler and the HANDIHALER inhaler in the corresponding treatment periods based on the randomisation scheme, and at the end of 2 periods, complete the inhaler preference questionnaire. Subjects will self-administer the inhalation once daily for 5-9 days in each treatment period.

This study will be placebo-only, and neither inhaler will contain active treatment. Subjects will continue their current COPD medication(s) as prescribed, and will follow up with their regular physician for their COPD healthcare during the study.

Approximately 211 subjects will be enrolled in the study.

ELLIPTA is a trademark of the GlaxoSmithKline group of companies. HANDIHALER is a trademark of Boehringer Ingelheim International GmbH.

ELIGIBILITY:
Inclusion Criteria:

* >=40 years of age at Visit 1.
* Diagnosis of COPD with a documented history of COPD for at least 6 months.
* Severity of Disease: Post albuterol/salbutamol forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) ratio <0.70 and FEV1 <=70% of predicted obtained within two years of Visit 1.
* Smoking History: Current or former (defined as subjects who have quit smoking for at least 3 months prior to Screening/Visit 1) cigarette smokers with a >10 pack-year smoking history. Number of pack years = (number of cigarettes per day/20) x number of years smoked (for example, 10 pack-years is equal to 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years).
* Current COPD Therapy:

  1. Currently receiving maintenance therapy with one or more long-acting bronchodilators, such as a long-acting muscarinic antagonist (LAMA; also known as a long-acting anti-cholinergic), long-acting beta 2-agonist (LABA), or inhaled corticosteroid (ICS)/LABA combination for the treatment of COPD. Subjects must be able to continue using their currently prescribed COPD maintenance inhaler therapy throughout the study and as needed short acting beta-adrenergic agonist (SABA) or short acting muscarinic antagonist (SAMA) for rescue use.
  2. Has been on current maintenance COPD treatment for at least 4 weeks prior to Screening/Visit 1 and evaluated as unlikely to change COPD treatment within 4 weeks of Visit 1.
* Males or
* Females who are not pregnant or not planning a pregnancy during the study or not lactating.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions defined for this study.
* Subject understands and is willing, able, and likely to comply with study procedures and restrictions.
* Subject must be able to read, comprehend, and record information in English.

Exclusion Criteria:

* Asthma: Subjects with a current diagnosis of asthma. Subjects with a prior history of asthma are eligible if they have a current diagnosis of COPD.
* Recent experience with the ELLIPTA inhaler: Subjects who used any ELLIPTA inhaler within 6 months (180 days) prior to Visit 1.
* Recent experience with the HANDIHALER inhaler: Subjects who used any HANDIHALER inhaler within 6 months (180 days) prior to Visit 1.
* Poorly controlled COPD: Subjects with symptoms of poorly controlled COPD such as:

  1. Acute worsening of COPD that is managed by the subject with corticosteroids or antibiotics or that requires treatment prescribed by a physician, in the 4 weeks prior to Visit 1.
  2. Hospitalization due to acute worsening of COPD within 4 weeks of Visit 1.
  3. Use of a total of 8 puffs/day or more of short-acting symptom relief medications such as albuterol and ipratropium for 2 consecutive days or any 3 days within 7 days immediately preceding Visit 1.
  4. Changes in COPD symptoms and signs, suggesting worsening COPD health status at Visit 1.
* Other Disease Abnormalities:

  1. Subjects with suspected or evidence of oropharyngeal candidiasis.
  2. Historical or current evidence of clinically significant or rapidly progressing or unstable cardiovascular, neurological, renal, hepatic, immunological, endocrine (including uncontrolled diabetes or thyroid disease) or haematological abnormalities that are uncontrolled. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which would affect the analysis if the disease/condition exacerbated during the study.
  3. Subjects with a history of psychiatric disease, intellectual deficiency, poor motivation or other conditions that will limit the validity of informed consent to participate in the study.
* Compliance: Subjects at risk of non-compliance, or unable to comply with the study procedures, or unable to continue their current COPD medications.
* Drug/alcohol abuse: Subjects with a known or suspected alcohol or drug abuse at Visit 1 which in the opinion of the investigator could interfere with the subject's proper completion of the protocol requirement.
* Drug/Food Allergy: A history of hypersensitivity to any components of the study inhaler (for example, lactose, magnesium stearate). In addition, subjects with a history of severe milk protein allergy that, in the opinion of the study physician, contraindicates participation will also be excluded.
* Investigational Product: Subjects who have received an investigational drug and/or medical device within 30 days of entry into this study (Screening/Visit 1), or within five drug half-lives of the investigational drug, whichever is longer.
* Affiliation with Investigator's Site: A subject will not be eligible for this study if he/she is an immediate family member of the participating investigator, sub-investigator, study coordinator, or employee of the participating investigator.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2016-06-21 (Actual); Primary Completion 2016-10-04 (Actual); Study Completion 2016-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (22):
- United States (22):
  - GSK Investigational Site, Glendale, Arizona
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Natchitoches, Louisiana
  - GSK Investigational Site, Sunset, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Plymouth, Minnesota
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Anderson, South Carolina
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Easley, South Carolina
  - GSK Investigational Site, Gaffney, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Rock Hill, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Union, South Carolina
  - GSK Investigational Site, Killeen, Texas
  - GSK Investigational Site, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Collison KA, Patel P, Preece AF, Stanford RH, Sharma RK, Feldman G. A Randomized Clinical Trial Comparing the ELLIPTA and HandiHaler Dry Powder Inhalers in Patients With COPD: Inhaler-Specific Attributes and Overall Patient Preference. COPD. 2018 Feb;15(1):46-50. doi: 10.1080/15412555.2017.1400000. Epub 2017 Dec 11. PMID 29227727
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants who met the inclusion criteria at screening were randomized to use ELLIPTA inhaler and Handihaler inhaler in a crossover manner at Visit 1 and Visit 2 once daily for 5-9 days. At Visit 3, participants were asked to complete the inhaler preference questionnaire.
Pre-assignment Details: A total of 227 participants with diagnosis and documented history of chronic obstructive pulmonary disease (COPD) were screened for this open-label, cross-over study, of which 13 were screen failures, 2 were randomized by error and did not receive treatment and 212 participants entered the study treatment phase.
Groups:
- ELLIPTA and HandiHaler: Participants were randomized to receive placebo using ELLIPTA inhaler and HandiHaler inhaler once daily for 5-9 days each in a crossover manner along with their routine COPD medication.
Period: Overall Study
Arm/Group | ELLIPTA and HandiHaler
Started | 212
Completed | 207
Not Completed | 5
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Arm/Group | ELLIPTA and HandiHaler
Number analyzed (Participants) | 212
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.1 (9.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 109
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: African American/African Heritage | 22
  Race/Ethnicity: American Indian or Alaska Native | 1
  Race/Ethnicity: Asian - Japanese Heritage | 1
  Race/Ethnicity: White - Arabic/North African Heritage | 1
  Race/Ethnicity: White - White/Caucasian/European Heritage | 187

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Preferring the Inhaler Based on the Number of Steps Needed to Take the COPD Medication
Description: Preference between ELLIPTA inhaler and Handihaler based on the number of steps needed to take the medication was assessed by the inhaler preference questionnaire at Visit 3 or Early Withdrawal (EW) visit. The responses were analyzed using a Cochran-Mantel-Haenszel test, adjusted for study inhaler use sequence and preference questionnaire version. The analysis was performed on the Modified Intent-to-treat (ITT) Population comprised of all participants in the ITT Population (comprised all randomized participants who received 1 dose of at least 1 study inhaler) who completed at least one question from the 5 preference questions.
Time Frame: Up to 18 days
Population: Modified ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | ELLIPTA and HandiHaler
Number analyzed (Participants) | 208
Percentage of participants
  ELLIPTA inhaler | 73
  HandiHaler | 20
  No preference | 7
Statistical Analysis 1: Comparison: ELLIPTA and HandiHaler; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel

2. Secondary Outcome: Percentage of Participants Preferring the Inhaler Based on How Easy it Was to Tell How Many Doses Were Left
Description: Preference between ELLIPTA inhaler and Handihaler based on how easy it was to tell how many doses were left was assessed by the inhaler preference questionnaire at Visit 3 or EW visit. The responses were analyzed using a Cochran-Mantel-Haenszel test, adjusted for study inhaler use sequence and preference questionnaire version.
Time Frame: Up to 18 days
Population: Modified ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | ELLIPTA and HandiHaler
Number analyzed (Participants) | 208
Percentage of participants
  ELLIPTA inhaler | 70
  HandiHaler | 18
  No preference | 12
Statistical Analysis 1: Comparison: ELLIPTA and HandiHaler; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel

3. Secondary Outcome: Percentage of Participants Preferring the Inhaler Based on the Size of the Inhaler
Description: Preference between ELLIPTA inhaler and HandiHaler based on the size of the inhaler was assessed by the inhaler preference questionnaire at Visit 3 or EW visit. The responses were analyzed using a Cochran-Mantel-Haenszel test, adjusted for study inhaler use sequence and preference questionnaire version.
Time Frame: Up to 18 days
Population: Modified ITT Population
Measure: Number; unit: Percentage of participants
Arm/Group | ELLIPTA and HandiHaler
Number analyzed (Participants) | 208
Percentage of participants
  ELLIPTA inhaler | 52
  HandiHaler | 25
  No preference | 24
Statistical Analysis 1: Comparison: ELLIPTA and HandiHaler; Test type: Other; p < 0.001, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: On-treatment serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of the study treatment until the follow-up contact.
Description: AEs and SAEs were collected in ITT Population which comprised of all participants who have been randomized and received one dose from at least one study inhaler.
Groups:
- ELLIPTA: Participants received ELLIPTA inhaler at Visit 1/Visit 2 once daily for 5-9 days.
- HandiHaler: Participants received HandiHaler inhaler at Visit 1/ Visit 2 once daily for 5-9 days.
Arm/Group | ELLIPTA | HandiHaler
Serious Adverse Events (participants affected / at risk) | 0/208 | 2/212
Other Adverse Events (participants affected / at risk) | 0/208 | 0/212
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ELLIPTA (N=208) | HandiHaler (N=212)
Sepsis (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.